CLINICAL TRIAL: NCT04823806
Title: Autophagy Characterization and Multi-level Molecular Profiling of Spermidine Supplementation: a Clinical Study
Brief Title: An Exploratory Clinical Study on Autophagy and Multi-level Molecular Profiling During Spermidine Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Dr. Nils Gassen, Dr. rer. nat. Nils Gassen, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: StressLess
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Depression; Healthy
Keywords: Spermidine; Autophagy; Depression
MeSH Terms: conditions — Depression | interventions — Spermidine

STUDY DESIGN:
Intervention Model Description: 2 groups of different inclusion criteria (healthy or depressive disorder) each group undergoing one out of two conditions (spermidine vs. placebo Supplementation) (randomized)
Who Masked: Participant, Investigator
Masking Description: double-blind study (participants nor experimenters know who receives placebo or spermidine supplementation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy participants and participants with depressive disorder: dietary spermidine supplementation (Experimental): Dietary Supplement: Polyamine 21 days of spermidine supplementation (3 sachets/day = 6mg spermidine/day)
  Interventions: Dietary Supplement: Spermidine (spermidineLIFE ®) OR Placebo
- Healthy participants and participants with depressive disorder: dietary placebo supplementation (Placebo Comparator): Dietary Supplement: Placebo 21 days of Placebo supplementation (3 sachets/day)
  Interventions: Dietary Supplement: Spermidine (spermidineLIFE ®) OR Placebo

INTERVENTIONS:
Dietary Supplement: Spermidine (spermidineLIFE ®) OR Placebo — 21 day of 6mg spermidine OR Placebo supplementation per day

SUMMARY:
Recently, the autophagy inducing caloric restriction mimic spermidine became available. Autophagy is essential for energy and cellular homeostasis through protein catabolism and dysregulation results in compromised proteostasis, stress-coping behavior, and in excessive secretion of signaling molecules and inflammatory cytokines. Antidepressants for example effect autophagy dependent pathways to exert their beneficial effects. It can therefore be hypothesized that autophagy induction through spermidine supplementation also shows beneficial clinical effect, particularly in the field of psychiatric conditions. It would be safe, low cost and easy to implement in relay to psychotropic medication in the treatment of psychiatric patients.Therefore, the aim of the project is to analyze clinical effects of spermidine supplementation in correlation to the underlying, multi-level molecular profiling.

DETAILED DESCRIPTION:
Recently, the autophagy inducing caloric restriction mimic spermidine-rich wheat germ extract (spermidineLIFE ®, from here onwards: spermidine) was approved by the European Food Safety Authority (EFSA) and became commercially available for use. Spermidine is safe, well tolerated and as caloric restriction mimetic an easy alternative if fasting is too challenging, e.g. for psychiatric patients. Research on spermidine in animal models is limited, but a study with mice overexpressing spermidine/spermine N1-acetyltransferase (SSAT) an enzyme of spermidine catabolism, suggests that these mice may be more prone to stress. An association between spermidine supplementation and improved memory performance as well as reduced mortality has been shown in an epidemiological correlation. So far laboratory and molecular assessments are missing. It is therefore of great interest to perform broad multidisciplinary studies of behavioral changes with plasma spermidine levels, the quantification of autophagic flux, and protein acetylation levels as well as molecular signaling in a longitudinal fashion to establish an epidemiological triangulation between spermidine, autophagy and (mental) health.

This study is a monocentric, randomized, double-blind, placebo-controlled trial in which a 3-week spermidine-based nutritional supplementation (6 mg/d; target intervention) will be compared to 3-weeks of placebo administration (control intervention). Recruitment of 40 healthy individuals and 40 individuals with diagnosed depressive disorder is planned, who will be allocated to one of the two study arms (n = 20 per intervention). At different time points (baseline, intervention day 7, 14 and 21, as well as one week follow up after the last intervention day) serval psychometrical questionnaires will be gathered and blood will be collected. Sleep quality will be additionally assessed by actigraphy. At selected days blood will be collected. Following, autophagy activity will be assessed by Western Blot analysis, and mass spectrometry based proteomics, phosphoproteomics, metabolomics and lipidomics will be performed. Bioinformatic analysis, statistical evaluation, quality control, and in silico pathway analyses will then specifically identify factors and cascades of relevance. Furthermore it is of great interest, whether epigenetic changes take place during spermidine supplementation and whether these are stable throughout the follow up analysis.

The aim of the project is to analyze clinical effects of spermidine supplementation in correlation to the underlying, multi-level molecular profiling. Longitudinal multi-omic profiling including proteome, metabolome, lipidome, and epigenetic changes will reveal time-series analysis of thousands of molecular changes and an orchestrated composition of autophagy depended signaling. The resulting findings will advance the role of autophagy in the development of psychiatric disorders, investigate alternative treatment options on a molecular level, and finally contribute to a better clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Present written declaration of consent
* Healty or diagnosed with depression
* BMI between 17 and 40

Exclusion Criteria:

* Insufficient linguistic communication
* Pregnancy or lactation
* Gluten, histamine or wheat seedling intolerance
* Drug abuse or alcohol dependency
* Current spermidine substitution

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Proteomics and autophagy processes | change from baseline over 21 days of supplementation to 7 day follow up
  Change in protein levels of autophagy biomarkers (LC3II & p62) of isolated PBMCs (peripheral blood mononuclear cells) by Western Blotting.

SECONDARY OUTCOMES:
Epigenetic patterns | change from baseline to day 21 of supplementation to 7 day follow up
  Evaluate epigenetic methylation patterns through blood based epigenome analysis
Proteome/phosphoproteome/ubiquitinome patterns | change from baseline over 21 days of supplementation to 7 day follow up
  Change in protein levels and protein phosphorylation by untargeted mass spectrometry-based proteomics and phosphoproteomics of isolated PBMCs (peripheral blood mononuclear cells).
Metabolic processes | change from baseline over 21 days of supplementation to 7 day follow up
  Targeted and quantitative analysis by mass spectrometry of change in metabolites of Plasma.
Lipid profiling | change from baseline over 21 days of supplementation to 7 day follow up
  Targeted and quantitative analysis by mass spectrometry of change in plasma Lipids.
Exosomal protein patterns | change from baseline over 21 days of supplementation to 7 day follow up
  Evaluate exosomal protein content through mass spectrometry based analysis
Glomerular filtration rate | change from baseline over 21 days of supplementation to 7 day follow up
  Estimated glomerular filtration rate (eGFR) in milliliter per minute (mL/min)
Cystatin C | change from baseline over 21 days of supplementation to 7 day follow up
  Cystatin C in Milligram per Liter (mg/L)
Liver Enzymes | change from baseline over 21 days of supplementation to 7 day follow up
  Alanine transaminase (ALT) and aspartate transaminase (AST) (U/L)
White blood cell differential | change from baseline over 21 days of supplementation to 7 day follow up
  Absolute number (per Liter) and relative amounts of neutrophils, lymphocytes, monocytes, eosinophils, basophils, and immature granulocytes (in %)
Saliva Cortisol Levels (dexamethasone suppression test) | on day 19 and 20 of supplementation
  Comparison of Saliva Cortisol Levels in nmol per Liter (nmol/L) after Dexamethason intake between spermidine and Placebo group
Sleep Efficiency | change from baseline over 21 days of supplementation to 7 day follow up
  Assessment of Sleep Efficiency (total time in bed/time asleep during night) by GenActive Aktigraphs
Overall sleep Quality | change from baseline over 21 days of supplementation to 7 day follow up
  Sleep diary to assess overall sleep quality assessed as ratio of the total time spent asleep (in hours) to the total amount of time spent in bed (in hours) per night
Sleep Quality (PSQI) | Change from baseline to day 7 day follow up visit
  Pittsburgh Sleep Quality Index (PSQI): self-report questionnaire to assess sleep quality over a 1-month time interval consisting of 19 individual items.
Mental well-being (WEMWBS) | Change from baseline to day 14 of supplementation to the 7 day follow up visit
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS): self-reported 14-item scale to assess Overall mental well-being
Resilience behavior (Wagnild &Young) | change from baseline over 21 days of supplementation to 7 day follow up
  Resilience scale (Wagnild &Young): self-reported 25-item scale to assess overall resilience
Spermidine blood concentration | change from baseline over 21 days of supplementation to 7 day follow up
  Assessment of spermidine blood Levels by HPLC (high pressure liquid chromatography) analysis
white cell count | change from baseline over 21 days of supplementation to 7 day follow up
  Complete white cell count (per liter)
Hemoglobin | change from baseline over 21 days of supplementation to 7 day follow up
  Hemoglobin (g/dL)
Hematocrit | change from baseline over 21 days of supplementation to 7 day follow up
  Hematocrit (%)
red cell count | change from baseline over 21 days of supplementation to 7 day follow up
  complete red cell count (per liter)
MCV | change from baseline over 21 days of supplementation to 7 day follow up
  mean corpuscular volume (fl)
MCH | change from baseline over 21 days of supplementation to 7 day follow up
  mean corpuscular hemoglobin (pg)
thrombocytes | change from baseline over 21 days of supplementation to 7 day follow up
  thrombocytes per Liter
MCHC | change from baseline over 21 days of supplementation to 7 day follow up
  mean corpuscular hemoglobin concentration (g/dL)
RDW | change from baseline over 21 days of supplementation to 7 day follow up
  red cell distribution width (%)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Clinic for psychiatry and psychotherapy, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eisenberg T, Knauer H, Schauer A, Buttner S, Ruckenstuhl C, Carmona-Gutierrez D, Ring J, Schroeder S, Magnes C, Antonacci L, Fussi H, Deszcz L, Hartl R, Schraml E, Criollo A, Megalou E, Weiskopf D, Laun P, Heeren G, Breitenbach M, Grubeck-Loebenstein B, Herker E, Fahrenkrog B, Frohlich KU, Sinner F, Tavernarakis N, Minois N, Kroemer G, Madeo F. Induction of autophagy by spermidine promotes longevity. Nat Cell Biol. 2009 Nov;11(11):1305-14. doi: 10.1038/ncb1975. Epub 2009 Oct 4. PMID 19801973
- [Result] Madeo F, Eisenberg T, Pietrocola F, Kroemer G. Spermidine in health and disease. Science. 2018 Jan 26;359(6374):eaan2788. doi: 10.1126/science.aan2788. PMID 29371440
- [Result] Fond G, Macgregor A, Leboyer M, Michalsen A. Fasting in mood disorders: neurobiology and effectiveness. A review of the literature. Psychiatry Res. 2013 Oct 30;209(3):253-8. doi: 10.1016/j.psychres.2012.12.018. Epub 2013 Jan 15. PMID 23332541
- [Result] Galluzzi L, Bravo-San Pedro JM, Levine B, Green DR, Kroemer G. Pharmacological modulation of autophagy: therapeutic potential and persisting obstacles. Nat Rev Drug Discov. 2017 Jul;16(7):487-511. doi: 10.1038/nrd.2017.22. Epub 2017 May 19. PMID 28529316
- [Result] Jia J, Le W. Molecular network of neuronal autophagy in the pathophysiology and treatment of depression. Neurosci Bull. 2015 Aug;31(4):427-34. doi: 10.1007/s12264-015-1548-2. Epub 2015 Aug 8. PMID 26254058